CLINICAL TRIAL: NCT02357706
Title: Comparison of Auto-Adjusting Positive Airway Pressure Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MA240115
Record Dates: First submitted 2015-01-27; First posted 2015-02-06 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 1) will use APAP A on the first night of the evaluation, and APAP B on the second night.
  Interventions: Device: APAP A (ResMed AirSense AutoSet); Device: APAP B (Apex iCH Auto)
- Group 2 (Active Comparator): Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 2) will use APAP B on the first night of the evaluation and APAP A on the second night.
  Interventions: Device: APAP A (ResMed AirSense AutoSet); Device: APAP B (Apex iCH Auto)

INTERVENTIONS:
Device: APAP A (ResMed AirSense AutoSet) — Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  Other Names: Auto-Adjusting Positive Airway Pressure Device A
Device: APAP B (Apex iCH Auto) — Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  Other Names: Auto-Adjusting Positive Airway Pressure Device B

SUMMARY:
Little is understood about how different auto-adjusting PAP devices operate. The purpose of this evaluation is to compare two devices in a randomised two night PSG trial.

ELIGIBILITY:
Inclusion Criteria:

* Males aged ≥ 18 years
* Recently diagnosed with OSA (AHI ≥15). Recently defined as less than 3 months before study entry
* Naive to CPAP therapy
* Participants willing and able to give written informed consent

Exclusion Criteria:

* Participants requiring Bi-level PAP
* Participants requiring supplemental oxygen
* Participants who are pregnant
* Subjects who have a pre existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Fietz, Prof, Principal Investigator — Charite Center of Sleep Medicine
Locations (1):
- Center of Sleep Medicine, Charité - Universitätsmedizin Berlin, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- APAP A, Then APAP B: Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 1) will use APAP A on the first night of the evaluation, and APAP B on the second night.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
- APAP B, Then APAP A: Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 2) will use APAP B on the first night of the evaluation and APAP A on the second night.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Period: Overall Study
Arm/Group | APAP A, Then APAP B | APAP B, Then APAP A
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Patients will be randomised to either "APAP A, then APAP B" or "APAP B, then APAP A". Patients in "APAP A, then APAP B" will use APAP A on the first night of the evaluation, and APAP B on the second night. Patients in "APAP B, then APAP A" will use APAP B on the first night of the evaluation and APAP A on the second night.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 31.1 (5.3)
Neck Size [Mean (Standard Deviation); unit: cm] | 41.1 (3.6)
waist-to-hip ratio [Mean (Standard Deviation); unit: ratio] | 1.01 (0.06)

OUTCOME MEASURES:

1. Primary Outcome: Mean Apnoea-Hypopnoea-Index (AHI)
Description: AHI measures the number of apnoeas + hypopnoeas per hours of night (events/hour).
Time Frame: 1 night (446 minutes) for APAP A (AirSense), 1 night (436 minutes) for APAP B (Apex)
Population: 20 patients have used APAP A, for which the primary outcome was calculated. The same 20 patients have used APAP B for which the Primary outcome was calculated.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- APAP A (AirSense Auto Set): Patients in the "APAP A, then APAP B" group (group 1) will use APAP A on the first night of the evaluation, and APAP B on the second night. Afterwards the outcome will be calculated for all 20 patients having used treatment APAP A.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
- APAP B (Apex iCH Auto): Patients in the "APAP B, then APAP A" group will use APAP B on the first night of the evaluation and APAP A on the second night. Afterwards the outcome will be calculated for all 20 patients having used treatment APAP A.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Arm/Group | APAP A (AirSense Auto Set) | APAP B (Apex iCH Auto)
Number analyzed (Participants) | 20 | 20
events/hour | 6.21 (6.73) | 7.45 (7.57)
Statistical Analysis 1: Comparison: APAP A (AirSense Auto Set) vs APAP B (Apex iCH Auto); Comparison of AHI/ oxygen desaturation index (ODI) of Device A compared with Device B. Efficacy is defined as a residual AHI and ODI on each night of the trial. PSG scored AHI and ODI will be collected on both trial nights (excluding the ramp period); and compared using the Paired T test; Test type: Non-Inferiority or Equivalence — We are testing the Hypothesis that there is a significant difference between CPAP A and CPAP B The Null Hypothesis is H0 = One CPAP is inferior to the other CPAP The Alternate Hypothesis is H1 = There is no significant difference between the CPAPs; p = 0.537, t-test, 1 sided; Mean Difference (Final Values) = 1.24
Statistical Analysis 2: Comparison: APAP A (AirSense Auto Set) vs APAP B (Apex iCH Auto); Test type: Non-Inferiority — We are testing the Hypothesis that there is a significant difference between CPAP A and CPAP B The Null Hypothesis is H0 = One CPAP is inferior to the other CPAP The Alternate Hypothesis is H1 = There is no significant difference between the CPAPs The expected difference mu is 0 events/hr The Non-Inferiority Margin delta is 0.75 events/hr (A difference of 1 event per hour is seen as clinically significant. 0.75 has been chosen to ensure any AHI change is seen); p = 0.05, t-test, 1 sided; Mean Difference (Net) = 1.24

2. Primary Outcome: Mean Oxygen Desaturation Index (ODI)
Description: Number of times that Oxygen Level Drops by 3% below baseline value, Events/hour
Time Frame: 1 night (446 minutes) for APAP A, 1 night (436 minutes) for APAP B.
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- APAP A (AirSense): Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 1) will use APAP A on the first night of the evaluation, and APAP B on the second night. Afterwards the outcome will be calculated for all 20 patients having used treatment APAP A.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
- APAP B (Apex): Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 2) will use APAP B on the first night of the evaluation and APAP A on the second night. Afterwards the outcome will be calculated for all 20 patients having used treatment APAP B.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
events/hour | 7.94 (8.10) | 10.63 (9.5)
Statistical Analysis 1: Comparison: APAP A (AirSense) vs APAP B (Apex); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.205, t-test, 1 sided; Mean Difference (Net) = 2.69
Statistical Analysis 2: Comparison: APAP A (AirSense) vs APAP B (Apex); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; p = 0.134, t-test, 1 sided; Mean Difference (Net) = 2.69

3. Secondary Outcome: Obstructive Apnoea Index (OAI)
Description: Number of obstructive apnoeas per hour of nights sleep, Events/hour
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
events/hour | 0.580 (1.525) | 0.885 (1.668)

4. Secondary Outcome: Central Apnoea Index (CAI)
Description: Number of central apnoeas during hours of sleep, events/hour
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- APAP B: Patients will be randomised to either Group 1 or Group 2. Patients in this group (group 2) will use APAP B on the first night of the evaluation and APAP A on the second night. Afterwards the outcome will be calculated for all 20 patients having used treatment APAP B.
  APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
  APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Arm/Group | APAP A (AirSense) | APAP B
Number analyzed (Participants) | 20 | 20
events/hour | 2.36 (4.08) | 2.51 (5.14)

5. Secondary Outcome: Mixed Apnoea Index (MAI)
Description: Number of obstructive and central apnoeas per hours of nights sleep, Events/hour
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
events/hour | 0.115 (0.514) | 0.220 (0.744)

6. Secondary Outcome: Hypopnoea-Index HI
Description: Number of Hypopnoeas per hour of nights sleep, Events/hour
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
events/hour | 3.17 (3.80) | 5.49 (5.51)

7. Secondary Outcome: Respiratory Effort Related Arousals RERAs
Description: Number of RERAs per hour of nights sleep, Events/hour
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
events/hour | 0.0 (0.0) | 2.81 (12.81)

8. Secondary Outcome: Flow Limitation (%)
Description: Percent of flow-limited breaths in relation to the overall breaths at night.
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: % overall breaths
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
% overall breaths | 49.25 (27.61) | 43.16 (22.59)

9. Secondary Outcome: Mean O2 Saturation
Description: Mean blood oxygen Saturation, %
Time Frame: 1 night (446 minutes) for APAP A; 1 night (436 minutes) for APAP B
Measure: Mean (Standard Deviation); unit: % total hemoglobin
Arm/Group | APAP A (AirSense) | APAP B (Apex)
Number analyzed (Participants) | 20 | 20
% total hemoglobin | 94.210 (2.414) | 93.680 (2.192)

ADVERSE EVENTS:
Groups:
- APAP A (AirSense): APAP A (ResMed AirSense AutoSet): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
- APAP B (Apex): APAP B (Apex iCH Auto): Commercially available device used to treat obstructive sleep apnea. The device automatically senses breathing and adjusts delivered pressure based on obstructive events
Arm/Group | APAP A (AirSense) | APAP B (Apex)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No